CLINICAL TRIAL: NCT07137884
Title: A Phase II, Multicenter, Randomized, Controlled Clinical Study of Anlotinib Hydrochloride Capsules as Maintenance Therapy for Intermediate-High Risk Rhabdomyosarcoma in Children
Brief Title: Anlotinib Hydrochloride Capsules in Maintenance Treatment for Intermediate-High Risk Rhabdomyosarcoma in Children
Acronym: ALTER-02
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Director, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-409-01
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Rhabdomyosarcoma Recurrent; Maintenance Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination medication group (Experimental)
  Interventions: Drug: Anlotinib+Cyclophosphamide+Vinorelbine
- Conventional maintenance treatment (Active Comparator)
  Interventions: Drug: Cyclophosphamide+Vinorelbine

INTERVENTIONS:
Drug: Anlotinib+Cyclophosphamide+Vinorelbine — Anlotinib hydrochloride capsules combined with Cyclophosphamide+Vinorelbine), Anlotinib hydrochloride capsules 8mg (weight ≤35kg) or 12mg (weight > 35kg), po, qd, D1-D14;on an empty stomach ,Two weeks off for one week，with a cycle of 3 weeks.
  Cyclophosphamide 25mg/m2, po, qd, D1-D28, with a cycle of 4 weeks. vinorelbine 60g/m2, po, qw, D1, 8,15, with a cycle of 4 weeks.
  Arms: Combination medication group
Drug: Cyclophosphamide+Vinorelbine — Cyclophosphamide 25mg/m2, po, qd, D1-D28, with a cycle of 4 weeks. vinorelbine 60mg/m2, po, qw, D1, 8,15, with a cycle of 4 weeks.
  Arms: Conventional maintenance treatment

SUMMARY:
This is a randomized controlled phase II clinical study aimed at evaluating the efficacy and safety of anlotinib hydrochloride in children with Intermediate-High -risk rhabdomyosarcoma. The study enrolled children with rhabdomyosarcoma confirmed by histopathology, with a clinical risk classification of high or Intermediate-risk accompanied by high-risk factors (high-risk factors are defined as age > 10 years，Poor prognosis molecular characteristics or those who cannot undergo surgery/radiotherapy);One year of maintenance treatment with anlotinib can increase the duration of response and long-term survival.

DETAILED DESCRIPTION:
Anlotinib Hydrochloride is a novel multi-target tyrosine kinase inhibitor.It can effectively inhibit kinases such as VEGFR, PDGFR, FGFR, c-Kit and Met, and has the functions of anti-tumor angiogenesis and inhibiting tumor growth.Especially for vascular endothelial growth factor receptor 2 (VEGFR2/KDR) and VEGFR3 shows a highly selective inhibitory effect, with a half-maximal inhibitory concentration (IC50) of less than 1.0 nM, which is significant, and has a significant anti-angiogenic effect.

ELIGIBILITY:
Inclusion Criteria:1.Age ≥5 years old, ≤18 years old, no gender restrictions; 2.ECOG performance status (PS) 0-3 points; 3.The expected survival period is not less than 12 weeks; 4.with high-risk or intermediate-risk rhabdomyosarcoma with high-risk factors (high-risk factors are defined as age > 10 years, poor prognostic molecular features, or inoperable/radiotherapy-ineligible) confirmed by histopathology ; 5.Complete remission was achieved after first-line treatment. 6.Patients must have fully recovered from the acute toxic effects of all prior anticancer chemotherapy: 7.Myelosuppressive chemotherapy: at least 21 days after the last myelosuppressive chemotherapy (42 days if nitrosoureas were used previously); 8.Investigational drugs or anticancer therapies other than chemotherapy: should not be used within the first 28 days of the planned start of anlotinib . Patients must have fully recovered from clinically significant toxicity of the therapy; 9.Hematopoietic growth factors: at least 14 days after the last dose of long-acting growth factors or 3 days after the last dose of short-acting growth factors; 10.Immunotherapy: at least 14 days after completing any type of immunotherapy (except steroids), such as immune checkpoint inhibitors and tumor vaccines; 11.X-ray therapy (XRT): at least 14 days after local palliative XRT (small-scale oral); if other parenchymal bone marrow (BM) irradiation is performed, including previous radioiodinated metaiodobenzylguanidine (131I-MIBG) treatment, it must be completed at least 42 days; 12.Stem cell infusion without total body irradiation (TBI): No evidence of active graft-versus-host disease, and the patient must have completed at least 56 days after transplantation or stem cell infusion; 13.Laboratory tests during the screening period should meet the following conditions: Absolute neutrophil count ( ANC) ≥ 1.5 × 109/L (ANC ≥ 1.0 × 109/L if bone marrow involvement occurs) Platelet count ( PLT) ≥75 × 109/L (PLT ≥50 × 109/L if bone marrow involvement occurs) Bilirubin ≤ 1.5 times ULN Creatinine ≤ 1.5 times ULN (calculated according to the standard Cockcroft-Gault formula) ALT/AST ≤ 3 times ULN (can be relaxed to 5 times ULN if liver metastasis is present) 14.Ability to comply with outpatient treatment, laboratory monitoring, and necessary clinical visits during study participation; 15.The parent/guardian of the child or adolescent subject is capable of understanding, agreeing to, and signing the Informed Consent Form (ICF) and applicable Child Assent Form before initiating any protocol-related procedures; and the subject is capable of expressing consent (where applicable) with the consent of the parent/guardian.

Exclusion Criteria:Patients with any of the following cannot be enrolled in this study :

1. Hypertensive patients who are currently receiving combined treatment with two or more antihypertensive drugs;
2. Patients with the following cardiovascular diseases: Myocardial ischemia or myocardial infarction of grade II or above, poorly controlled arrhythmia (including QTc interval ≥450 ms for men and ≥470 ms for women); Grade III to IV heart failure according to NYHA standards, or left ventricular ejection fraction (LVEF) <50% as indicated by cardiac ultrasound examination;
3. Patients with a history of or concurrent interstitial lung disease;
4. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 ULN), bleeding tendency or receiving thrombolytic or anticoagulant therapy;
5. Daily hemoptysis of two teaspoons or more before enrollment;
6. Patients with clinically significant bleeding symptoms or a clear bleeding tendency within 3 months prior to enrollment, such as gastrointestinal bleeding, bleeding hemorrhoids, bleeding gastric ulcers, baseline fecal occult blood ++ or above, or vasculitis;
7. Arterial/venous thrombotic events occurring within 12 months prior to enrollment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
8. Known hereditary or acquired bleeding and thrombotic tendencies (such as hemophilia, coagulation disorders, thrombocytopenia, hypersplenism, etc.);
9. Long-term unhealed wounds or fractures (pathological fractures caused by tumors are not included);
10. Patients who have undergone major surgery or suffered severe traumatic injury, fracture or ulcer within 4 weeks of enrollment;
11. Factors that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
12. Abdominal fistula, gastrointestinal perforation, or abdominal abscess within 6 months before enrollment ;
13. Urinalysis indicates urine protein ≥++, and the 24-hour urine protein volume is confirmed to be ≥1.0 g;
14. Serous cavity effusion (including pleural effusion, ascites, and pericardial effusion) with clinical symptoms requiring symptomatic treatment;
15. Note: Asymptomatic patients with serous cavity effusion can be enrolled. Patients with symptomatic serous cavity effusion who have undergone active symptomatic treatment (anti-cancer drugs cannot be used to treat serous cavity effusion) and are judged by the researchers to be eligible for enrollment are allowed to be enrolled.
16. Active infection requiring antimicrobial treatment (e.g., antibacterial drugs, antiviral drugs, excluding anti-hepatitis B treatment for chronic hepatitis B and antifungal drugs);
17. Those with a history of psychotropic drug abuse and unable to quit, or those with mental disorders;
18. Participated in other anti-tumor drug clinical trials within 4 weeks before enrollment;
19. Patients who have previously or concurrently suffered from other uncured malignant tumors, except for cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and superficial bladder cancer;
20. Use of drugs or foods that are known strong CYP3A4 inhibitors within 7 days before the first dose, including but not limited to: atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinafil, ritonavir, saquinavir, telithromycin, troleandomycin, and voriconazole;
21. Use of drugs known to be strong inducers of CYP3A4 within 12 days prior to the first dose, including but not limited to: carbamazepine, phenobarbital, phenytoin, rifabutin , and rifampicin;
22. Pregnant or breastfeeding women; patients of childbearing potential who are unwilling or unable to take effective contraceptive measures;
23. The researcher determines other situations that may affect the conduct of the clinical study and the determination of the study results.
24. When virological testing during the screening period shows any of the following:

HBsAg positive and HBV DNA above the upper limit of normal Anti-HCV positive and HCV RNA positive HIV positive

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
DOR (Duration of Response) | 2 year
  DOR (Duration of Response) refers to the period from the first assessment of complete response (CR) or partial response (PR) of the tumor to the first assessment of disease progression (PD) or death from any cause.

SECONDARY OUTCOMES:
2-year DFS rate | 2 year after treatment
  The 2-year DFS rate refers to the probability that a patient does not experience disease recurrence or progression within 2 years after cancer treatment.
2-year OS rate | 2 year after treatment
  2-year OS rate is defined as the percentage of patients who do not experience death from any cause after 2-year treatment.
Adverse events (AE) | 2 year
  An AE refers to any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, but which does not necessarily have a causal relationship with this treatment. Number and classification of participants with treatment-related adverse events as assessed by CTCAE v5.0 were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Gongdong, China